CLINICAL TRIAL: NCT04778670
Title: Artificial Intelligence in a Population-based Breast Cancer Screening - the Prospective Clinical Trial ScreenTrust CAD
Brief Title: Artificial Intelligence in Large-scale Breast Cancer Screening
Acronym: ScreenTrustCAD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Capio Sankt Görans Hospital (Other); Lunit Inc. (Industry); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Fredrik Strand, Registrar (biträdande överläkare), Karolinska University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Triple | Purpose: Diagnostic
Other Study IDs: STGKS001; EPM 2020-00487 (Other: Ethical Review Authority (Sweden)); K 2020-0807 (Other: Karolinska University Hospital)
Record Dates: First submitted 2021-02-22; First posted 2021-03-03 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Breast Neoplasm Female
Keywords: Artificial Intelligence; Breast Cancer; Mammography; Screening
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective clinical trial following a paired screen-positive design (Pepe, Alonzo; 2001), with the aims to assess the performance of an AI algorithm combined with radiologists(s) compared to standard-of-care being two radiologists assessing screening mammograms in a true screening population. Since all decisions by individual readers will be recorded, it is possible to determine what the outcome would have been had one or two of the readers not been allowed to assess images, and to determine what the outcome would have been had the recall decision been performed by consensus decision (actual) compared to single reader arbitration of discordant cases.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Positive disease status is ascertained by pathology-verified breast cancer. Disease status is not known to any of the actors (except for the outcomes assessor by necessity). AI decision is not known by the care provider radiologists until they have made their decisions. In the subsequent consensus discussion where a decision is made to recall or not to recall a woman, the AI decision is known. After AI decision has been recorded and outcomes have been assessed, the investigators will have full information on outcomes and AI decisions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care means all examinations will receive a flagging decision by: first reader and second reader radiologist as usual. However, in this paired design all participants will belong to both arms.
  Interventions: Diagnostic Test: Radiologist reading
- AI CAD combination (Experimental): AI CAD combination in the primary end-point means the combination of the flagging decision of the first reader and AI CAD; in the secondary end-points it means any combination of AI alone, or AI in combination with first, second and both readers.
  Interventions: Diagnostic Test: AI CAD; Diagnostic Test: Radiologist reading

INTERVENTIONS:
Diagnostic Test: AI CAD — The Lunit INSIGHT MMG will be used as the AI CAD in our study. Initially, version 1.6.1.1 will be installed. The software version will be continuously updated with subsequent software releases, after confirming in a historic calibration dataset that the performance is improved. The operating point will be set based on a historic calibration dataset to attain a joint sensitivity of breast cancer detection of AI and first reader which is 2% higher than for first and second reader.
  Other Names: Lunit INSIGHT MMG
  Arms: AI CAD combination
Diagnostic Test: Radiologist reading — Standard of care, each radiologist will assess the mammography examination, making a binary flagging decision (flag the examination to continue to consensus discussion, or not)

SUMMARY:
This is a prospective clinical trial following a paired screen-positive design, with the aims to assess the performance of an artificial intelligence (AI) computer-aided detection (CAD) algorithm as an independent reader, in addition to two radiologists, of screening mammograms in a true screening population. Since all decisions by individual readers will be recorded, it is possible to determine what the outcome would have been had one or two of the readers not been allowed to assess images, and to determine what the outcome would have been had the recall decision been performed by consensus decision (actual) compared to single reader arbitration of discordant cases.

ELIGIBILITY:
Inclusion Criteria:

* Participants in regular population-based breast cancer screening at Capio St Göran Hospital

Exclusion Criteria:

* Incomplete exam (complete exam: mediolateral oblique and craniocaudal images of Left and Right breast)
* Breast implant
* Complete mastectomy (excluded from screening positive group)
* Participant in surveillance program for prior breast cancer

Ages: 40 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55579 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incident breast cancer | At Screening
  Breast cancer diagnosis by pathologist
Incident breast cancer | Within 12 months after screening
  Breast cancer diagnosis by pathologist
Incident breast cancer | Within 23 months after screening
  Breast cancer diagnosis by pathologist

SECONDARY OUTCOMES:
Reader flagging | At screening
  Radiologist or AICAD assessing the mammograms as suspicious or not suspicious for malignancy
Consensus recall | At screening
  A decision by the consensus discussion to recall the woman for further work-up
Tissue sampling | At screening
  Biopsy or fine needle aspiration performed
Process failure | At screening
  Failure of the AI CAD software to generate AI scores

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Strand, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Capio St Göran Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
To the extent allowed by source institution, legal agreements, and applicable laws and regulations
Supporting Information: Study Protocol, SAP
Time Frame: At study start
Access Criteria: Anyone can access study protocol and SAP.

REFERENCES:
- [Derived] Dembrower KE, Crippa A, Eklund M, Strand F. Human-AI Interaction in the ScreenTrustCAD Trial: Recall Proportion and Positive Predictive Value Related to Screening Mammograms Flagged by AI CAD versus a Human Reader. Radiology. 2025 Mar;314(3):e242566. doi: 10.1148/radiol.242566. PMID 40100021
- [Derived] Dembrower K, Crippa A, Colon E, Eklund M, Strand F; ScreenTrustCAD Trial Consortium. Artificial intelligence for breast cancer detection in screening mammography in Sweden: a prospective, population-based, paired-reader, non-inferiority study. Lancet Digit Health. 2023 Oct;5(10):e703-e711. doi: 10.1016/S2589-7500(23)00153-X. Epub 2023 Sep 8. PMID 37690911

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-05-16): https://cdn.clinicaltrials.gov/large-docs/70/NCT04778670/Prot_SAP_002.pdf